CLINICAL TRIAL: NCT02946268
Title: Up-down Sequential Allocation Study to Determine the Optimal Volume, Rate, and Interval of Bolus of Ropivacaine 0.2% in Interscalene Continuous Nerve Catheters for Shoulder Surgery
Brief Title: Optimal Volume, Rate, and Interval of Bolus Nerve Catheters for Shoulder Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00072762
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2018-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Volume of bolus (Experimental): Ropivacaine 0.2% volume increased or decreased by 1ml based on previous patient experience. If pain greater than or equal to 5/10 in the previous patient, the current patient will receive an increase in volume of bolus by 1ml. If pain is less than 5/10 in the previous patient the current patient will receive a decrease in volume by 1ml.
  Interventions: Drug: Ropivacaine
- Rate of delivery of bolus (Experimental): Ropivacaine 0.2% rate increased or decreased by 50ml/hr based on previous patient experience. If pain greater than or equal to 5/10 in the previous patient at 30 minutes, the current patient will receive an increase in rate of bolus by 50ml/hr. If the pain is less than 5/10 the rate will be decreased by 50ml/hr.
  Interventions: Drug: Ropivacaine
- Interval between bolus (Experimental): Ropivacaine 0.2% interval increased or decreased by 1 hour based on previous patient experience. If the previous patient received pain score of 2/10 at 2 hours then the current patient will have an interval of three hours. If the pain is greater than 2/10, the interval will be shortened by 1 hour.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Change in administration of ropivacaine. Rate, Volume and Interval of bolus altered.
  Other Names: Naropin

SUMMARY:
The purpose of this study is to determine the ideal delivery of local anesthetics for pain control when using continuous interscalene peripheral nerve catheters for shoulder surgery.

The study will be conducted in three stages. In the first stage the ideal bolus volume of ropivacaine will be determined. In the second stage the optimal rate of delivery of the bolus (infusion rate) will be determined. Finally, once both the ideal volume and infusion rate has been determined, the optimal interval between boluses of local anesthetic will be determined.

DETAILED DESCRIPTION:
The purpose of this study is to determine the ideal delivery of local anesthetics for postoperative analgesia when using continuous interscalene peripheral nerve catheters for shoulder surgery. New technology has emerged with electronic pumps that permit intermittent mandatory boluses of local anesthetic to be delivered in addition to continuous infusions. The pump would automatically deliver a bolus at a given interval, but would otherwise be idle for a period of time. This technology could improve the efficacy of local anesthetics, and thereby improve postoperative analgesia.

Continuous peripheral nerve catheters have been shown to improve pain control in several orthopedic surgical procedures when compared to opioids. However, it is not uncommon for patients to experience breakthrough pain in spite of a functional peripheral nerve block. Many times, this breakthrough pain can be managed with a bolus of local anesthetic administered by an anesthesia provider. Until recently, the vast majority of peripheral nerve catheter infusion pumps have only had the capability of providing a constant rate of local anesthetic administration. Newer technology allows for infusion pumps to deliver intermittent mandatory boluses of local anesthetic. This technique of local anesthetic administration has previously been evaluated with popliteal nerve blocks, but to our knowledge has never been evaluated for use with interscalene nerve catheters.

Currently, data would support the idea that a bolus of local anesthetic can improve analgesia with decreased side effects compared to a continuous infusion. However, there is little data evaluating the optimal volume of bolus, the optimal speed of delivery, or the optimal interval between local anesthetic boluses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years of age
* Patients scheduled to undergo unilateral shoulder surgery at Duke University Medical Center, including arthroscopic rotator cuff repair, acromioplasty, hemiarthroplasty, and total shoulder replacement.
* American Society of Anesthesiology (ASA) Physical Class 1-3.
* BMI ≤40 kg/m2

Exclusion Criteria:

* Patients with a contraindication to placement of interscalene nerve block. This includes abnormal clotting, skin infection involving the neck, the presence of neurological disorders or cervical spine disease, contralateral phrenic nerve dysfunction, or moderate-severe COPD (FEV1<80% of normal values and/or FEV1/FVC < 0.70)
* Patients with chronic pain (pain existing for longer than 6 months), or taking chronic opioids (greater than 60 morphine equivalents per day) at time of surgery
* Contraindications to or known drug interactions with local anesthetics
* Patients who will be discharged home directly from PACU
* Planned administration of another investigational product or procedure during the subject's participation in this study.
* Patients who do not have the capacity to give legally effective consent
* Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postoperative course.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Optimal Volume of Ropivacaine 0.2% bolus via interscalene catheter | 1 day
  Up-down sequential allocation alteration of volume to determine optimal volume of bolus

SECONDARY OUTCOMES:
Optimal Rate of Ropivacaine 0.2% administration bolus via interscalene cathter | 1 day
  Up-down sequential allocation alteration of rate to determine optimal rate of bolus

OTHER OUTCOMES:
Optimal Interval of Ropivacaine 0.2% administration of bolus via interscalene catheter | 1 day
  Up-down sequential allocation alteration of interval to determine optimal interval of bolus

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Dooley, MD, Principal Investigator — Duke University
Locations (1):
- Duke Ambulatory Surgery Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No